CLINICAL TRIAL: NCT03427177
Title: Mychoice: Testing an Interactive mHealth Tool to Enhance Communication and Informed Decision Making About Clinical Trial Participation in Cancer Patients
Brief Title: Mychoice: Testing an Interactive mHealth Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); University of Pennsylvania (Other); Temple University (Other); Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17-8013
Record Dates: First submitted 2017-11-21; First posted 2018-02-09 (Actual); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2020-12

CONDITIONS: Conflict; Decisional Conflict

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants randomized to the treatment arm of the study will be given the mychoice tool.
  Interventions: Behavioral: mychoice
- Control (No Intervention): Participants randomized to the control arm of the study will be given existing literature from the NCI that describes clinical trials (standard information for newly diagnosed cancer patients).

INTERVENTIONS:
Behavioral: mychoice — The mychoice communication tool begins to prepare patients to participate in a personal and tailored discussion with their provider about clinical trials as a potential treatment option. It is also customized to address the concerns of those least likely to participate, instead of providing a more general look at clinical trials- a common trait of other available tools.
  Arms: Treatment

SUMMARY:
Investigators aim to test a culturally diverse and patient guided mHealth decision tool called mychoice, which allows patients to explore their concerns and questions related to clinical trial participation, as well as create a customized and personalized set of questions to enhance patient-provider communication and increase informed decision making. This study employs a mixed-methods approach using both qualitative and quantitative data to evaluate the effectiveness of the mychoice intervention for patients and to explore the provider and organizational factors that impact implementation. A randomized controlled trial will be performed with 270 participants in order to determine the acceptability and feasibility of the intervention, as well as its effects on self-efficacy in discussing clinical trial participation with providers, leading to enhanced informed decision-making. A secondary aim of the study is to evaluate the implementation of the intervention in clinical settings. Implementation evaluation will occur using surveys of medical staff whose patients are participating in the study. These surveys will assess institutional facilitators and barriers to study implementation. Investigators will also conduct cognitive de-briefing interviews after the intervention is completed with key stakeholders at the participating institutions, which will inform a larger implementation study in the future.

DETAILED DESCRIPTION:
Evidence shows that although clinical trials are aimed at producing new strategies for reducing cancer morbidity and mortality, participation remains sub-optimal for all populations, especially those from racial and ethnic groups. Although some interventions have been found to be effective at enhancing participation, few studies have tested tailored communication activities using innovative communication techniques (perceptual mapping) with aims to address barriers and facilitators for patients and facilitate more engaged discussions with their providers in real world settings.

Participation in clinical trials is a serious and complex decision, and many patients of all races and backgrounds have limited knowledge and understanding of clinical trials as a treatment option. Although research has been conducted to explore the barriers to participation, there has been a call for more intervention research to address these barriers. A fundamental aspect of patient focused interventions is an exploration of their personal questions and concerns, without which it is difficult for patients to become empowered to participate in an informed or shared decision making process. However, there remains limited empirical research to suggest which messages are most salient to a diverse range of patients to improve decision making, and how decision tools can be tailored to enhance patient-provider communication. This research will provide insight into that process when the decision is participation in clinical trials.

Evidence shows that ethnic and racial minorities are significantly underrepresented in clinical trials, which is critical to producing new strategies for reducing cancer morbidity and mortality for all populations. Recognizing the complexity of barriers to participation in clinical trials, research has focused on potential strategies to enhance participation. Interventions have shown that provider referrals of minority patients, community outreach, acknowledging and addressing issues of trust, flexibility in intervention methods, and population targeted materials are effective. Few studies, however, have tested tailored communication activities to address barriers and facilitators for patients using innovative communication techniques in real world settings - meaning ways these activities can be integrated into the healthcare workflow - or addressed the unique needs of racial and ethnic minorities.

The mychoice communication tool begins to prepare patients to participate in a personal and tailored discussion with their provider about clinical trials as a potential treatment option. The tool is also customized to address the concerns of those least likely to participate, instead of providing a more general look at clinical trials- a common trait of other available tools. Previous research has shown that patient education before the first oncologist visit improves knowledge, attitudes, and preparation for decision making about clinical trials and integrating these tools into the clinical encounter is critical. In addition, using innovative communication techniques (perceptual mapping and vector modeling) to validate and explore notable messages across diverse cancer patients provided new insights into tailoring messages and personalizing patient/provider communication. Insight gained from validation of the intervention will improve the decision making process and inform a large scale integration of mychoice to affect patient perceptions and increase willingness to participate in clinical trials, especially in minority patients.

In addition, Investigators will assess barriers to implementation when introducing the tool in diverse cancer centers, each with different protocols and patient populations, to inform a future proposal. Using the Consolidated Framework for Implementation Science (CFIR), one of the predominant implementation science research frameworks, we will focus on five domains: intervention characteristics, outer settings, inner setting, characteristics of individuals (patients and providers), and process. Implementation science is becoming an important component of intervention implementation and we aim to use this framework to ensure success.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* Active diagnosis of invasive cancer (any diagnoses), pre or post chemo/radiation/surgery
* Able to speak and read English

Exclusion Criteria:

* Participated in a therapeutic trial in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Fleisher, PhD, Principal Investigator — Fox Chase Cancer Center; Sarah Bass, PhD, Principal Investigator — Temple
Locations (5):
- United States (5):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Temple University Health System, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Baquet CR, Henderson K, Commiskey P, Morrow JN. Clinical trials: the art of enrollment. Semin Oncol Nurs. 2008 Nov;24(4):262-9. doi: 10.1016/j.soncn.2008.08.006. PMID 19000600
- [Background] Comis R, Crowley J. Baseline study of patient accrual onto publically sponsored U.S. cancer clinical trials: an analysis conducted for the global access project of the national patient advocate foundation, 2006.
- [Background] Michaels, M.S., S; ENACCT and Community-Campus Partnerships for Health, Communities as Partners in Cancer Clinical Trials: Changing Research, Practice and Policy. 2008: Silver Springs, MD.
- [Background] Weinberg, A.D. Eliminating Disparities in Clinical Trials. cited 2009 June 4th, 2009; Version 2: Available from: http://www.bcm.edu/edict/home.html.
- [Background] Colon-Otero G, Smallridge RC, Solberg LA Jr, Keith TD, Woodward TA, Willis FB, Dunn AN. Disparities in participation in cancer clinical trials in the United States : a symptom of a healthcare system in crisis. Cancer. 2008 Feb 1;112(3):447-54. doi: 10.1002/cncr.23201. PMID 18085590
- [Background] Gadegbeku CA, Stillman PK, Huffman MD, Jackson JS, Kusek JW, Jamerson KA. Factors associated with enrollment of African Americans into a clinical trial: results from the African American study of kidney disease and hypertension. Contemp Clin Trials. 2008 Nov;29(6):837-42. doi: 10.1016/j.cct.2008.06.001. Epub 2008 Jun 27. PMID 18639652
- [Background] Katz RV, Wang MQ, Green BL, Kressin NR, Claudio C, Russell SL, Sommervil C. Participation in biomedical research studies and cancer screenings: perceptions of risks to minorities compared with whites. Cancer Control. 2008 Oct;15(4):344-51. doi: 10.1177/107327480801500409. PMID 18813202
- [Background] Shavers VL, Lynch CF, Burmeister LF. Factors that influence African-Americans' willingness to participate in medical research studies. Cancer. 2001 Jan 1;91(1 Suppl):233-6. doi: 10.1002/1097-0142(20010101)91:1+3.0.co;2-8. PMID 11148585
- [Background] Mills EJ, Seely D, Rachlis B, Griffith L, Wu P, Wilson K, Ellis P, Wright JR. Barriers to participation in clinical trials of cancer: a meta-analysis and systematic review of patient-reported factors. Lancet Oncol. 2006 Feb;7(2):141-8. doi: 10.1016/S1470-2045(06)70576-9. PMID 16455478
- [Background] Todd AM, Laird BJ, Boyle D, Boyd AC, Colvin LA, Fallon MT. A systematic review examining the literature on attitudes of patients with advanced cancer toward research. J Pain Symptom Manage. 2009 Jun;37(6):1078-85. doi: 10.1016/j.jpainsymman.2008.07.009. Epub 2009 May 5. PMID 19419837
- [Background] Evelyn B, Toigo T, Banks D, Pohl D, Gray K, Robins B, Ernat J. Participation of racial/ethnic groups in clinical trials and race-related labeling: a review of new molecular entities approved 1995-1999. J Natl Med Assoc. 2001 Dec;93(12 Suppl):18S-24S. PMID 11798060
- [Background] Stewart JH, Bertoni AG, Staten JL, Levine EA, Gross CP. Participation in surgical oncology clinical trials: gender-, race/ethnicity-, and age-based disparities. Ann Surg Oncol. 2007 Dec;14(12):3328-34. doi: 10.1245/s10434-007-9500-y. Epub 2007 Aug 8. PMID 17682824
- [Background] Rivera-Goba MV, Dominguez DC, Stoll P, Grady C, Ramos C, Mican JM. Exploring decision-making of HIV-infected Hispanics and African Americans participating in clinical trials. J Assoc Nurses AIDS Care. 2011 Jul-Aug;22(4):295-306. doi: 10.1016/j.jana.2010.10.007. Epub 2011 Jan 21. PMID 21256054
- [Background] Symonds RP, Lord K, Mitchell AJ, Raghavan D. Recruitment of ethnic minorities into cancer clinical trials: experience from the front lines. Br J Cancer. 2012 Sep 25;107(7):1017-21. doi: 10.1038/bjc.2012.240. Epub 2012 May 31. PMID 23011540
- [Background] Schmotzer GL. Barriers and facilitators to participation of minorities in clinical trials. Ethn Dis. 2012 Spring;22(2):226-30. PMID 22764647
- [Background] Advani AS, Atkeson B, Brown CL, Peterson BL, Fish L, Johnson JL, Gockerman JP, Gautier M. Barriers to the participation of African-American patients with cancer in clinical trials: a pilot study. Cancer. 2003 Mar 15;97(6):1499-506. doi: 10.1002/cncr.11213. PMID 12627515
- [Background] Goldberg D. The case for Eliminating Disparities in Clinical Trials. J Cancer Educ. 2009;24(2 Suppl):S34-8. doi: 10.1007/BF03182310. No abstract available. PMID 20024824
- [Background] Gross CP. Racial disparities in clinical trial enrolment. Lancet. 2008 Nov 15;372(9651):1713-4. doi: 10.1016/S0140-6736(08)61714-6. No abstract available. PMID 19013309
- [Background] Newman LA, Roff NK, Weinberg AD. Cancer clinical trials accrual: missed opportunities to address disparities and missed opportunities to improve outcomes for all. Ann Surg Oncol. 2008 Jul;15(7):1818-9. doi: 10.1245/s10434-008-9869-2. Epub 2008 Apr 19. No abstract available. PMID 18425554
- [Background] Ford JG, Howerton MW, Lai GY, Gary TL, Bolen S, Gibbons MC, Tilburt J, Baffi C, Tanpitukpongse TP, Wilson RF, Powe NR, Bass EB. Barriers to recruiting underrepresented populations to cancer clinical trials: a systematic review. Cancer. 2008 Jan 15;112(2):228-42. doi: 10.1002/cncr.23157. PMID 18008363
- [Background] Gul RB, Ali PA. Clinical trials: the challenge of recruitment and retention of participants. J Clin Nurs. 2010 Jan;19(1-2):227-33. doi: 10.1111/j.1365-2702.2009.03041.x. PMID 20500260
- [Background] Markman M, Petersen J, Montgomery R. An examination of the influence of patient race and ethnicity on expressed interest in learning about cancer clinical trials. J Cancer Res Clin Oncol. 2008 Jan;134(1):115-8. doi: 10.1007/s00432-007-0263-4. Epub 2007 Jun 28. PMID 17598129
- [Background] Adderley-Kelly B, Green PM. Strategies for successful conduct of research with low-income African American populations. Nurs Outlook. 2005 May-Jun;53(3):147-52. doi: 10.1016/j.outlook.2005.03.004. PMID 15988452
- [Background] Knobf MT, Juarez G, Lee SY, Sun V, Sun Y, Haozous E. Challenges and strategies in recruitment of ethnically diverse populations for cancer nursing research. Oncol Nurs Forum. 2007 Nov;34(6):1187-94. doi: 10.1188/07.ONF.1187-1194. PMID 18024345
- [Background] Lai GY, Gary TL, Tilburt J, Bolen S, Baffi C, Wilson RF, Howerton MW, Gibbons MC, Tanpitukpongse TP, Powe NR, Bass EB, Ford JG. Effectiveness of strategies to recruit underrepresented populations into cancer clinical trials. Clin Trials. 2006;3(2):133-41. doi: 10.1191/1740774506cn143oa. PMID 16773955
- [Background] Davis SW, Fleisher L, Ter Maat J, Muha C, Laepke K. Treatment and clinical trials decisionmaking: the impact of the Cancer Information Service. Part 5. J Health Commun. 1998;3 Suppl:71-85. doi: 10.1080/108107398127265. PMID 10977271
- [Background] Meropol NJ, Wong YN, Albrecht T, Manne S, Miller SM, Flamm AL, Benson AB 3rd, Buzaglo J, Collins M, Egleston B, Fleisher L, Katz M, Kinzy TG, Liu TM, Margevicius S, Miller DM, Poole D, Roach N, Ross E, Schluchter MD. Randomized Trial of a Web-Based Intervention to Address Barriers to Clinical Trials. J Clin Oncol. 2016 Feb 10;34(5):469-78. doi: 10.1200/JCO.2015.63.2257. Epub 2015 Dec 23. PMID 26700123
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Denicoff AM, McCaskill-Stevens W, Grubbs SS, Bruinooge SS, Comis RL, Devine P, Dilts DM, Duff ME, Ford JG, Joffe S, Schapira L, Weinfurt KP, Michaels M, Raghavan D, Richmond ES, Zon R, Albrecht TL, Bookman MA, Dowlati A, Enos RA, Fouad MN, Good M, Hicks WJ, Loehrer PJ Sr, Lyss AP, Wolff SN, Wujcik DM, Meropol NJ. The National Cancer Institute-American Society of Clinical Oncology Cancer Trial Accrual Symposium: summary and recommendations. J Oncol Pract. 2013 Nov;9(6):267-76. doi: 10.1200/JOP.2013.001119. Epub 2013 Oct 15. PMID 24130252
- [Background] Maly RC, Frank JC, Marshall GN, DiMatteo MR, Reuben DB. Perceived efficacy in patient-physician interactions (PEPPI): validation of an instrument in older persons. J Am Geriatr Soc. 1998 Jul;46(7):889-94. doi: 10.1111/j.1532-5415.1998.tb02725.x. PMID 9670878
- [Background] Bennett C, Graham ID, Kristjansson E, Kearing SA, Clay KF, O'Connor AM. Validation of a preparation for decision making scale. Patient Educ Couns. 2010 Jan;78(1):130-3. doi: 10.1016/j.pec.2009.05.012. Epub 2009 Jun 26. PMID 19560303
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] Kriston L, Scholl I, Holzel L, Simon D, Loh A, Harter M. The 9-item Shared Decision Making Questionnaire (SDM-Q-9). Development and psychometric properties in a primary care sample. Patient Educ Couns. 2010 Jul;80(1):94-9. doi: 10.1016/j.pec.2009.09.034. Epub 2009 Oct 30. PMID 19879711
- [Background] Barr PJ, Thompson R, Walsh T, Grande SW, Ozanne EM, Elwyn G. Correction: the psychometric properties of CollaboRATE: a fast and frugal patient-reported measure of the shared decision-making process. J Med Internet Res. 2015 Feb 6;17(2):e32. doi: 10.2196/jmir.4272. No abstract available. PMID 25667387
- [Background] National Institutes for Health (NIH). NIH Demographics form Version 2.0.
- [Background] NCI's Health and Information National Trend Study. Computer Facility. PIES Study (Diefenbach et al)
- [Background] Morris NS, MacLean CD, Chew LD, Littenberg B. The Single Item Literacy Screener: evaluation of a brief instrument to identify limited reading ability. BMC Fam Pract. 2006 Mar 24;7:21. doi: 10.1186/1471-2296-7-21. PMID 16563164
- [Background] Hoerger M, Chapman BP, Mohile SG, Duberstein PR. Development and psychometric evaluation of the Decisional Engagement Scale (DES-10): A patient-reported psychosocial survey for quality cancer care. Psychol Assess. 2016 Sep;28(9):1087-100. doi: 10.1037/pas0000294. PMID 27537003

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 125 | 132
Completed | 92 | 105
Not Completed | 33 | 27

BASELINE CHARACTERISTICS:
Population: The number of participants in the Baseline Analysis Population only includes participants who completed the baseline survey in it's entirety. 257 participants were consented and joined the study; however, they did not complete any study tasks and no data was completed at baseline. 250 participants completed baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 122 | 128 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 68 | 81 | 149
  >=65 years | 54 | 47 | 101
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 79 | 158
  Male | 43 | 49 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 14
  Not Hispanic or Latino | 101 | 102 | 203
  Unknown or Not Reported | 16 | 17 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 45 | 50 | 95
  White | 68 | 68 | 136
  More than one race | 7 | 3 | 10
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 122 | 128 | 250

OUTCOME MEASURES:

1. Primary Outcome: Perceived Efficacy in Patient-Physician Interactions (PEPPI) Self-Efficacy Scale- Outcome Measure at Baseline, Post-test and One Month Follow-up
Description: 10-item scale measuring patient confidence in communicating with their physician. Participants respond to each question on a scale of 1 to 5, with 5 representing "very confident,'' and 1 representing "not at all confident." The range of possible scores for the full PEPPI scale is 10 to 50 (50 representing highest patient-perceived self-efficacy).
Time Frame: Baseline and post-test (both occur on same day, day 1), one month follow-up
Population: There was participant drop off between baseline, post-test, and follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 121 | 126
score on a scale
  Baseline | 44.6 (5.8) | 44.0 (8.3)
  Post-test: number analyzed (Participants) | 101 | 118
  Post-test | 44.3 (6.5) | 44.4 (7.1)
  Follow-up | 44.8 (6.0) | 44.2 (6.3)

2. Secondary Outcome: CollaboRATE Perceived Shared Decision Making Scale
Description: Measure of patient perceptions of physician effort to discuss concerns, 3 items. There is a possible range of 0-9 for each item.
  Higher scores represent more shared decision making.
Time Frame: 1 month follow-up
Population: Participants were only asked these questions if their doctor talked to them about participating in a clinical trial prior to completing follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 33 | 35
score on a scale
  How much effort was made to help you understand clinical trials? | 3.82 (1.185) | 3.74 (1.039)
  How much effort was made to listen to the things that matter most to you about clinical trials? | 3.76 (1.300) | 3.71 (1.017)
  How much effort was made to include what matters most to you in choosing what to do next? | 3.97 (1.185) | 3.69 (1.022)

3. Secondary Outcome: Shared Decision Making (SDM Q-9) Scale
Description: Measure of patient perception of shared decision making with provider (12 items). The instrument's statements are rated on a six-point scale from ''completely disagree'' (0) to ''completely agree'' (5).
  Higher means indicate higher levels of perceived shared decision making.
Time Frame: 1 month follow-up
Population: Only participants who were offered a clinical trial were asked these questions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 32 | 36
score on a scale
  My doctor made it clear that a decision needs to be made.: number analyzed (Participants) | 31 | 35
  My doctor made it clear that a decision needs to be made. | 4.19 (1.642) | 4.09 (1.652)
  My doctor wanted to know exactly how I want to be involved in making a decision.: number analyzed (Participants) | 31 | 35
  My doctor wanted to know exactly how I want to be involved in making a decision. | 4.29 (1.657) | 4.23 (1.592)
  My doctor toldme that there are different options for treating my medical condition. | 4.78 (1.237) | 4.67 (1.414)
  My doctor precisely explained the advantages and disadvantages of clinical trials.: number analyzed (Participants) | 32 | 35
  My doctor precisely explained the advantages and disadvantages of clinical trials. | 4.13 (1.755) | 4.20 (1.623)
  My doctor helped me understand all the information for clinical trials.: number analyzed (Participants) | 31 | 35
  My doctor helped me understand all the information for clinical trials. | 3.90 (1.578) | 4.29 (1.526)
  My doctor asked me which treatment option I prefer.: number analyzed (Participants) | 32 | 35
  My doctor asked me which treatment option I prefer. | 4.16 (1.798) | 4.49 (1.541)
  My doctor and I thoroughly weighed the different treatment options.: number analyzed (Participants) | 32 | 35
  My doctor and I thoroughly weighed the different treatment options. | 4.19 (1.857) | 4.69 (1.367)
  My doctor and I selected a treatment option together.: number analyzed (Participants) | 32 | 35
  My doctor and I selected a treatment option together. | 4.66 (1.619) | 4.54 (1.540)
  My doctor and I reached an agreement on how to proceed.: number analyzed (Participants) | 32 | 35
  My doctor and I reached an agreement on how to proceed. | 4.81 (1.52) | 4.60 (.479)

4. Secondary Outcome: Ottawa Decisional Conflict
Description: 13 item measure to determine patient clarity on the risks and benefits of clinical trials, support from friends and family, and patient decision regarding cancer treatment. Items are given a score value of: 0= 'strongly agree'; 2= 'neither agree nor disagree'; 3= 'disagree'; 4= 'strongly disagree' TOTAL SCORE 16 items [items 1-16 are inclusive] are: a) summed; b) divided by 16; and c) multiplied by 25. Scores range from 0 [no decisional conflict] to 100 [extremely high decisional conflict]
Time Frame: Baseline and post-test (both occur on same day, day 1), one month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 122 | 128
score on a scale
  Baseline | 32.0 (19.8) | 31.6 (20.5)
  Post-test | 24.5 (147) | 26.2 (18.8)
  Follow-up | 27.1 (18.3) | 28.7 (17.5)

5. Secondary Outcome: Preparation for Decision Making (PrepDM) Scale
Description: Measures preparedness of patient to make a decision (10 items) on a 1 "not at all" to 5 "a great deal" scale.
  Higher means indicated higher perceived level of preparation for decision making.
Time Frame: Post test (day 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 104 | 120
score on a scale
  How much did the edu... Help you recognize that a decision needs to be made about clinical trials? | 3.7 (1.1) | 3.7 (1.2)
  Prepare you to make a better decision about clinical trials? | 3.9 (.9) | 3.9 (1.1)
  Help you think about the pros and cons of treatment options? | 3.9 (1.0) | 3.9 (1.1)
  Help you think about which pros and cons are most important? | 3.9 (1.0) | 3.8 (1.2)
  Help you know that the decision depends on what matters most to you? | 4.1 (.9) | 4.0 (1.0)
  Help you organize your own thoughts about the decision? | 4.0 (1.0) | 3.9 (1.0)
  Help you think about how involved you want to be in this decision? | 4.1 (1.0) | 4.1 (1.0)
  Help you identify questions you want to ask your doctor? | 4.1 (.9) | 4.1 (1.0)
  Prepare you to talk to your doctor about what matters most to you? | 4.1 (.9) | 4.1 (1.0)
  Prepare you for a follow-up visit with your doctor? | 3.8 (1.0) | 3.9 (1.2)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between baseline and one-month follow-up.
Description: This was a minimal risk study.
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/128
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/128
Other Adverse Events (participants affected / at risk) | 0/122 | 0/128

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT03427177/Prot_SAP_000.pdf